CLINICAL TRIAL: NCT00420277
Title: A Randomized, Double-Blind, Phase III Study of the Efficacy and Safety of an Oxygen-Carrying Plasma Expander, Hemospan®, Compared With Voluven® toTreat Hypotension in Patients Undergoing Primary Hip Arthroplasty With Spinal Anesthesia
Brief Title: Phase III Study of Hemospan® for Treating Hypotension in Hip Arthroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6090
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Hypotension; Ischemia
Keywords: Hip arthroplasty; Anesthesia, spinal; Hypotension; Ischemia; Blood substitutes; Plasma expanders
MeSH Terms: conditions — Hypotension; Ischemia | interventions — maleimide-polyethylene glycol-modified hemoglobin, MP4; HES 130-0.4; Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hemospan (MP4OX) (Experimental): 4.3 g/dL MalPEG-Hb solution
  Interventions: Drug: Hemospan (MP4OX)
- Control (Active Comparator): Voluven (HES 130/0.4)
  Interventions: Drug: Voluven (HES 130/0.4)

INTERVENTIONS:
Drug: Hemospan (MP4OX) — 250 mL unit dose, up to 500 mL total dose as needed at protocol-defined dosing triggers
  Other Names: MP4OX solution; 4.3 g/dL MalPEG-Hb; PEGylated Hb
  Arms: Hemospan (MP4OX)
Drug: Voluven (HES 130/0.4) — 250 mL unit dose, up to 500 mL total dose as needed at protocol-defined dosing triggers
  Other Names: 6% HES 130/0.4; 6% hetastarch solution; Voluven
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether Hemospan is superior to Voluven for treatment of hypotensive episodes during the perioperative period (from induction of spinal anesthesia until 6 hours after skin closure), and for reducing the incidence of operative and postoperative complications including organ dysfunction and failure until follow-up at one month following surgery. An independent Data Safety Monitoring Board (DSMB) will periodically evaluate the safety data collected during this trial

DETAILED DESCRIPTION:
Hemospan is a novel hemoglobin-based oxygen carrier developed to perfuse and oxygenate tissue at risk for ischemia and hypoxia. As a result of its molecular size and oxygen binding characteristics, Hemospan selectively off-loads oxygen in tissues predisposed to low oxygen tension. Preclinical evidence suggests that Hemospan provides rapid and effective plasma expansion and tissue perfusion, and that the properties of Hemospan target oxygen release in the microcirculation.

Spinal anesthesia is the preferred choice for hip arthroplasty procedures in elderly patients, but is associated with a functional hypovolemia due to loss of vascular tone that frequently causes acute hypotensive episodes. Hypotension represents a surrogate marker of hypovolemia that may be further exacerbated by surgical bleeding, which can result in decreased cardiac output, insufficient perfusion and inadequate tissue oxygenation. Ischemia resulting from hypotension can adversely affect vital organ function and may result in complications and postoperative morbidity. As the population ages and more patients become candidates for orthopedic reconstruction or joint replacement surgery, the number of patients at risk is increasing. The ideal IV solution for treating hypovolemia-associated hypotension and improving hemodynamic stability would be an effective plasma expander that promotes tissue perfusion and delivers oxygen to ischemic or marginally hypoxic tissue.

Preclinical animal studies have shown that Hemospan may be well-suited to this application and may even be better than blood in some situations. Data from Sangart's Phase II orthopedic surgery study (No. 6055), published recently by Olofsson et al. (Anesthesiology 2006; 105(6):1153-63) support the safety and potential benefit of Hemospan for preventing and treating hypotension in orthopedic surgery patients undergoing hip replacement surgery under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective primary hip arthroplasty (based on an osteoarthritis diagnosis) under spinal anesthesia
* Adult male or female (surgically sterile or post-menopausal), aged 50 years or older
* American Society of Anesthesiology (ASA) Class II or III
* Physical examination, laboratory status, vital signs, and ECG within acceptable limits for the planned surgery, as judged by the investigator
* Have been given written and verbal information by the investigator about Hemospan and the protocol, and have had the opportunity to ask questions about the study
* Patients must sign an Informed Consent form that has been reviewed and approved by the independent Ethics Committee

Exclusion Criteria:

* Hip fracture patients and nail/pin extraction procedures
* Clinical evidence of uncontrolled cardiovascular, infectious, psychiatric, metabolic or systemic disorders including diabetes and rheumatoid arthritis
* Evidence of significant hypertension with SBP >180 mmHg, or a difference in SBP obtained in each arm that is >15 mmHg (measured in the supine position in both arms, at screening)
* Recent history or evidence of MI or stroke (within 6 months)
* Known alcohol or drug dependency
* Currently taking oral anti-coagulant therapy; except for low-dose aspirin (acetylsalicylic acid), <200 mg/day
* History of coagulopathy
* Involved in any investigational drug or device trial within 30 days prior to this study
* Professional or ancillary personnel involved with this study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Total duration of all hypotensive episodes occurring during anesthesia/surgery and throughout the postoperative period (defined as the first 6 hours following skin closure) | Up to 6 hours after skin closure

SECONDARY OUTCOMES:
Incidence of serious operative and postoperative complications, combined into a Composite Morbidity Outcome that includes acute heart failure, acute MI, ischemic stroke, and renal failure | 30 days
Incidence of operative and postoperative organ dysfunction related to ischemia and/or tissue hypoxia, as a Composite Ischemia Outcome that includes clinical evidence of cerebral ischemia, myocardial ischemia, and renal dysfunction | 30 days
Mortality (In-hospital, and all-cause at 30 days) | 30 days
Time to resolve/correct the initial hypotensive episode that led to the first dosing trigger | Intraoperative
Time to the second dosing trigger from the first dosing trigger | Intraoperative
Proportion of patients treated successfully with one dose | Intraoperative
Incidence of hypotension | Up to 6 hours after skin closure
Duration of the longest period of hypotension recorded | Up to 6 hours after skin closure
Incidence of intervention with a pressor agent to treat hypotensive episodes | Up to 6 hours after skin closure
Incidence of postoperative intervention with a diuretic for volume-overload or inadequate urine output | Post-operative day 3

CONTACTS AND LOCATIONS:
Overall Officials: Philippe van der Linden, MD, PhD, Principal Investigator — CHU Brugmann, Brussels
Locations (22):
- Belgium (3):
  - CHU Brugmann, Brussels
  - Z.O.L. Genk, Genk
  - Stedelijk Ziekenhuis Roeselare, Roeselare
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Motol, I. Ortopedicka klinika, Prague
  - Fakultni nemocnice Motol, II. Ortopedicka klinika, Prague
  - Fakultni nemocnice Na Bulovce, Prague
- Netherlands (4):
  - Medisch Spectrum Twente, Enschede
  - Tergooi Ziekenhuizen, locatie Hilversum, Hilversum
  - Sint Maartenskliniek, Nijmegen
  - UMC Erasmus, Rotterdam
- Poland (5):
  - Samodzielny Publiczny Szpital Kliniczny AM, Bialystok
  - SP Wojewódzki Szpital Chirurgii Urazowej, Piekary Śląskie
  - Wojewódzki Szpital Specjalistyczny nr 5, Sosnowiec
  - Instytut Reumatologii, Klinika Reumoortopedii, Warsaw
  - SK Dzieciątka Jezus, Warsaw
- Sweden (6):
  - Länssjukhuset Gävle, Gävle
  - Kalmar Hospital, Kalmar
  - Lasarettet Motala, Motala
  - Danderyd Sjukhus, Stockholm
  - Söder Hospital, Stockholm
  - Uddevalla Sjukhus, Uddevalla

REFERENCES:
- [Background] Bjorkholm M, Fagrell B, Przybelski R, Winslow N, Young M, Winslow RM. A phase I single blind clinical trial of a new oxygen transport agent (MP4), human hemoglobin modified with maleimide-activated polyethylene glycol. Haematologica. 2005 Apr;90(4):505-15. PMID 15820947
- [Background] Cabrales P, Tsai AG, Winslow RM, Intaglietta M. Effects of extreme hemodilution with hemoglobin-based O2 carriers on microvascular pressure. Am J Physiol Heart Circ Physiol. 2005 May;288(5):H2146-53. doi: 10.1152/ajpheart.00749.2004. Epub 2005 Jan 6. PMID 15637119
- [Background] Young MA, Riddez L, Kjellstrom BT, Bursell J, Winslow F, Lohman J, Winslow RM. MalPEG-hemoglobin (MP4) improves hemodynamics, acid-base status, and survival after uncontrolled hemorrhage in anesthetized swine. Crit Care Med. 2005 Aug;33(8):1794-804. doi: 10.1097/01.ccm.0000172648.55309.13. PMID 16096458
- [Background] Tsai AG, Cabrales P, Manjula BN, Acharya SA, Winslow RM, Intaglietta M. Dissociation of local nitric oxide concentration and vasoconstriction in the presence of cell-free hemoglobin oxygen carriers. Blood. 2006 Nov 15;108(10):3603-10. doi: 10.1182/blood-2006-02-005272. Epub 2006 Jul 20. PMID 16857991
- [Background] Winslow RM. Current status of oxygen carriers ('blood substitutes'): 2006. Vox Sang. 2006 Aug;91(2):102-10. doi: 10.1111/j.1423-0410.2006.00789.x. PMID 16907870
- [Background] Olofsson C, Ahl T, Johansson T, Larsson S, Nellgard P, Ponzer S, Fagrell B, Przybelski R, Keipert P, Winslow N, Winslow RM. A multicenter clinical study of the safety and activity of maleimide-polyethylene glycol-modified Hemoglobin (Hemospan) in patients undergoing major orthopedic surgery. Anesthesiology. 2006 Dec;105(6):1153-63. doi: 10.1097/00000542-200612000-00015. PMID 17122578
- [Background] Winslow RM. Red cell substitutes. Semin Hematol. 2007 Jan;44(1):51-9. doi: 10.1053/j.seminhematol.2006.09.013. PMID 17198847
- [Result] van der Linden P, Gazdzik TS, Jahoda D, Heylen RJ, Skowronski JC, Pellar D, Kofranek I, Gorecki AZ, Fagrell B, Keipert PE, Hardiman YJ, Levy H; 6090 Study Investigators. A double-blind, randomized, multicenter study of MP4OX for treatment of perioperative hypotension in patients undergoing primary hip arthroplasty under spinal anesthesia. Anesth Analg. 2011 Apr;112(4):759-73. doi: 10.1213/ANE.0b013e31820c7b5f. Epub 2011 Feb 11. PMID 21317165
- See also: Click here for more information about Sangart, Inc. — http://www.sangart.com